CLINICAL TRIAL: NCT00179361
Title: Natural History of Oral Cancer Precursors
Brief Title: Natural History of Oro-pharyngeal Cancer Precursors
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Nicolas Schlecht, PhD, Ass. Prof. Epidemiology & Population Health, Albert Einstein College of Medicine
Other Study IDs: 2003-434; DE016089-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Precancerous Conditions; Leukoplakia; Erythroplasia; Oral Papillomas
MeSH Terms: conditions — Precancerous Conditions; Leukoplakia; Erythroplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oral brush samples.
Oversight: Data Monitoring Committee: No

SUMMARY:
Oro-pharyngeal cancers can develop from squamous dysplastic precursor lesions, which occur in a subset of common white (leukoplakia), red (erythroplasia), or mixed oro-pharyngeal plaques. Known risk factors for oro-pharyngeal cancer include tobacco smoke, alcohol consumption, diet and, in a subset of tumors, human papillomavirus (HPV). Along the oro-pharyngeal disease continuum, there may be variations in gene expression precursor lesions as a result of exposure to smoking, alcohol and HPV. However, the components of gene expression that are most likely associated with tumorigenesis in these tissues are poorly understood. This study will focus upon early gene expression profiles in the oral cavity and oropharynx in subjects who have precursor lesions and have been exposed to the common risk factors for carcinoma development including smoking and HPV infection. This application is to conduct pilot testing and establish appropriate procedures for an international prospective cohort study of the natural history of oro-pharyngeal cancer precursors among men and women at high risk of oro-pharyngeal cancer at Montefiore Medical Center, Bronx-NY. Brush biopsy specimens will be used to collect a transepithelial sample of cells from oro-pharyngeal plaques, as well as normal tissue from defined regions of the oral and pharyngeal mucosa. Measurement of gene expression will employ novel high-throughput cDNA microarray analysis and PCR-based HPV DNA testing. Oro-pharyngeal dysplasia will be diagnosed using cytopathology. Under this application, we will assess our planned instruments and procedures on an initial sample of 40 subjects. This planning period will allow for precise identification of methodologies, standardization of instruments and assays to be utilized by additional participating centers in a subsequent application.

ELIGIBILITY:
Inclusion Criteria:

* Established residence in the greater Metropolitan area of New York City, including Westchester, Long Island, Southern Connecticut and Northern New Jersey

Exclusion Criteria:

* No history of therapy for oral cancer in the previous 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care Dental and Otolaryngology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2004-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas F Schlecht, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Result] Muller K, Kazimiroff J, Fatahzadeh M, Smith RV, Wiltz M, Polanco J, Grossberg RM, Belbin TJ, Strickler HD, Burk RD, Schlecht NF. Oral Human Papillomavirus Infection and Oral Lesions in HIV-Positive and HIV-Negative Dental Patients. J Infect Dis. 2015 Sep 1;212(5):760-8. doi: 10.1093/infdis/jiv080. Epub 2015 Feb 13. PMID 25681375